CLINICAL TRIAL: NCT02400333
Title: An Open-label, Randomised, Four-period, Four-treatment, Crossover, Single-centre, Single-dose Study to Assess the Bioavailability of Ticagrelor Orodispersible Tablets, Compared to Ticagrelor Immediate-release Tablets in Healthy Subjects
Brief Title: Study to Assess the Bioavailability of Ticagrelor OD Tablet vs. IR Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D5139C00003
Record Dates: First submitted 2015-03-09; First posted 2015-03-27 (Estimated); Results first posted 2016-08-03 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-08

CONDITIONS: Bioavailability; Healthy Subjects
Keywords: ticagrelor orodispersible tablet; ticagrelor immediate-release tablet; relative bioavailability; Phase I; healthy subjects
MeSH Terms: interventions — Water; Excipients; Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatments A-D-B-C sequence (Experimental): Treatment A in Period 1, Treatment D in Period 2, Treatment B in Period 3 and Treatment C in Period 4
  Interventions: Drug: Ticagrelor OD tablet (90 mg single dose) administered with 200 ml of water; Drug: Ticagrelor OD tablet (90 mg single dose) administered without water; Drug: Ticagrelor OD tablet (90 mg single dose) suspended in water administered via nasogastric tube; Drug: Brilique®, Ticagrelor IR tablet (90 mg) administered with 200mL of water
- Treatments B-A-C-D sequence (Experimental): Treatment B in Period 1, Treatment A in Period 2, Treatment C in Period 3 and Treatment D in Period 4
  Interventions: Drug: Ticagrelor OD tablet (90 mg single dose) administered with 200 ml of water; Drug: Ticagrelor OD tablet (90 mg single dose) administered without water; Drug: Ticagrelor OD tablet (90 mg single dose) suspended in water administered via nasogastric tube; Drug: Brilique®, Ticagrelor IR tablet (90 mg) administered with 200mL of water
- Treatments C-B-D-A sequence (Experimental): Treatment C in Period 1, Treatment B in Period 2, Treatment D in Period 3 and Treatment A in Period 4
  Interventions: Drug: Ticagrelor OD tablet (90 mg single dose) administered with 200 ml of water; Drug: Ticagrelor OD tablet (90 mg single dose) administered without water; Drug: Ticagrelor OD tablet (90 mg single dose) suspended in water administered via nasogastric tube; Drug: Brilique®, Ticagrelor IR tablet (90 mg) administered with 200mL of water
- Treatments D-C-A-B sequence (Experimental): Treatment D in Period 1, Treatment C in Period 2, Treatment A in Period 3 and Treatment B in Period 4
  Interventions: Drug: Ticagrelor OD tablet (90 mg single dose) administered with 200 ml of water; Drug: Ticagrelor OD tablet (90 mg single dose) administered without water; Drug: Ticagrelor OD tablet (90 mg single dose) suspended in water administered via nasogastric tube; Drug: Brilique®, Ticagrelor IR tablet (90 mg) administered with 200mL of water

INTERVENTIONS:
Drug: Ticagrelor OD tablet (90 mg single dose) administered with 200 ml of water — 90 mg single dose
  Other Names: Treatment A
Drug: Ticagrelor OD tablet (90 mg single dose) administered without water — 90 mg single dose
  Other Names: Treatment B
Drug: Ticagrelor OD tablet (90 mg single dose) suspended in water administered via nasogastric tube — 90 mg single dose
  Other Names: Treatment C
Drug: Brilique®, Ticagrelor IR tablet (90 mg) administered with 200mL of water — 90 mg single dose
  Other Names: Treatment D

SUMMARY:
This study will be an open-label, randomised, four-period, four-treatment, crossover study in healthy male and female of non-childbearing potential subjects, performed at a single study centre.

The objective of the study is to assess the bioavailability of ticagrelor orodispersible (OD) tablets when administered with water, without water and suspended in water to be administered through nasogastric tubes, compared to ticagrelor immediate-release (IR) tablets

DETAILED DESCRIPTION:
Study to evaluate the bioavailability of ticagrelor OD tablets administered with water, without water and suspended in water to be administered through nasogastric tubes, compared to ticagrelor IR tablets.

ELIGIBILITY:
Inclusion Criteria:

Healthy male and female subjects aged 18 to 55 years with suitable veins for cannulation or repeated venepuncture. - Females must have a negative pregnancy test at screening and on each admission to the clinical unit, must not be lactating, and must be of non-childbearing potential, confirmed at screening by fulfilling one of the following criteria: Postmenopausal defined as amenorrhoea for at least 12 months or more following cessation of all exogenous hormonal treatments and follicle-stimulating hormone (FSH) levels in the postmenopausal range or Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation. - Have a body mass index (BMI) between 18.5 and 29.9 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive. -Able to understand, read and speak the German language.

Exclusion Criteria: - History of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the potential subject at risk because of participation in the study, or influence the results or the potential subject's ability to participate in the study.

* Any abnormalities in alkaline phosphatase (ALP), alanine aminotransferase (ALT), aspartate aminotransferase (AST), gamma-glutamyl transpeptidase (GGT), urea, creatinine, thyroid-stimulating hormone (TSH), International Normalised Ratio (INR), activated partial thromboplastin time (aPTT), white blood cell (WBC) count, haemoglobin (Hb) or platelet count. Any other abnormal haematology, clinical chemistry, coagulation or urinalysis results, as judged with an unacceptable deviation that is considered to be clinically significant by the investigator.
* Any clinically significant abnormal findings in vital signs, as judged by the investigator. at screening and at baseline (Day -1 of Treatment period 1), defined as:

  * Systolic blood pressure < 90mmHg or ≥ 140 mmHg
  * Diastolic blood pressure < 50mmHg or ≥ 90 mmHg
  * Pulse < 50 or > 85 beats per minute (bpm)
* Current smokers or those who have smoked or used nicotine products within the previous 3 months.
* History of haemophilia, von Willebrand's disease, lupus anticoagulant, or other diseases/syndromes that can either alter or increase the propensity for bleeding.
* A personal history of vascular abnormalities including aneurysms; a personal history of severe haemorrhage, hematemesis, melena, haemoptysis, severe epistaxis, severe thrombocytopenia, intracranial haemorrhage; or rectal bleeding within 1 year prior to screening; or history suggestive of peptic ulcer disease; or at the discretion of the investigator.
* History of a clinically significant non-traumatic bleed or clinically significant bleeding risk, as judged by the investigator.
* Use of aspirin, ibuprofen, non-steroidal anti-inflammatory drugs (NSAIDs), or any other drug known to increase the propensity for bleeding for 2 weeks before randomisation.
* Platelet count less than 150 x 109/L.

Criteria applicable to insertion of a nasogastric tube:

* History of severe midface trauma and/or recent nasal surgery.
* History of coagulation abnormality, oesophageal varices or stricture, recent banding or cautery of oesophageal varices, and/or alkaline ingestion, at the discretion of the investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2015-06; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rainard Fuhr, Dr. med., Principal Investigator — PAREXEL International GmbH, Berlin
Locations (1):
- Research Site, Berlin, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at PAREXEL International, Early Phase Clinical Unit Berlin, Berlin, Germany. In this study, 100 participants were screened, out of which 36 were randomized and treated.
Pre-assignment Details: Participants were randomized in 4 sequence Williams design for 4 periods and 4 treatments:Ticagrelor orodispersible (OD) tablets with water (Treatment A);Ticagrelor OD tablets without water (Treatment B);Ticagrelor OD tablets suspended in water through nasogastric tube (Treatment C);Ticagrelor immediate-release (IR) tablets with water(Treatment D).
Groups:
- ADBC Sequence: Treatment A in Period 1, Treatment D in Period 2, Treatment B in Period 3 and Treatment C in Period 4.
- BACD Sequence: Treatment B in Period 1, Treatment A in Period 2, Treatment C in Period 3 and Treatment D in Period 4.
- CBDA Sequence: Treatment C in Period 1, Treatment B in Period 2, Treatment D in Period 3 and Treatment A in Period 4.
- DCAB Sequence: Treatment D in Period 1, Treatment C in Period 2, Treatment A in Period 3 and Treatment B in Period 4.
Period: Overall Study
Arm/Group | ADBC Sequence | BACD Sequence | CBDA Sequence | DCAB Sequence
Started | 9 | 9 | 9 | 9
Completed | 8 | 8 | 7 | 7
Not Completed | 1 | 1 | 2 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1
Not completed — Protocol Violation | 1 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ADBC Sequence | BACD Sequence | CBDA Sequence | DCAB Sequence | Total
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (12) | 44 (12) | 42 (13) | 40 (13) | 42 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 1 | 4
  Male | 8 | 8 | 8 | 8 | 32

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Ticagrelor and Its Active Metabolite AR-C124910XX.
Description: Blood samples for the determination of plasma concentrations of both ticagrelor and AR-C124910XX were collected at pre-dose (0 hours) and post-dose at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36 and 48 hours (14 samples per treatment period).
Time Frame: 0 hours (pre-dose) and post-dose at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36 and 48 hours in each treatment period.
Population: The Pharmacokinetic (PK) analysis set consisted of all participants in the safety analysis set for whom at least one of the primary PK parameters, for a given analyte, can be calculated for at least two treatment periods and who had no major protocol deviations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Treatment A: Participants received Ticagrelor OD tablets administered with water. The OD tablet was placed on the tongue to disintegrate and be swallowed subsequently with 200 mL noncarbonated water at room temperature.
- Treatment B: Participants received Ticagrelor OD tablets administered without water. The OD tablet was placed on the tongue to disintegrate and be swallowed subsequently with saliva.
- Treatment C: Participants received Ticagrelor OD tablets suspended in water to be administered through a nasogastric tube (NG) tube into the stomach (total of 200 mL of water).
- Treatment D: Participants received Ticagrelor IR tablets administered orally with 200 mL of water.
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 30 | 31 | 33 | 33
ng/mL
  Ticagrelor | 428 (25.0) | 499 (34.0) | 479 (32.1) | 520 (29.0)
  AR-C124910XX | 118 (26.5) | 126 (24.7) | 126 (30.4) | 129 (31.8)
Statistical Analysis 1: Comparison: Treatment A vs Treatment D; Statistical assessment of ticagrelor relative bioavailability following ticagrelor OD tablets administered with water compared to ticagrelor IR tablets; Test type: Superiority or Other; Geometric mean ratio = 84.85, 90% CI 2-sided [76.77 to 93.78]
Statistical Analysis 2: Comparison: Treatment B vs Treatment D; Statistical assessment of ticagrelor relative bioavailability following ticagrelor OD tablets administered without water compared to ticagrelor IR tablets; Test type: Superiority or Other; Geometric mean ratio = 96.61, 95% CI 2-sided [88.22 to 105.79]
Statistical Analysis 3: Comparison: Treatment C vs Treatment D; Statistical assessment of ticagrelor relative bioavailability following ticagrelor OD tablets suspended in water and administered through NG tube compared to ticagrelor IR tablets; Test type: Superiority or Other; Geometric mean ratio = 92.16, 95% CI 2-sided [85.59 to 99.25]
Statistical Analysis 4: Comparison: Treatment A vs Treatment D; Statistical assessment of metabolite AR-C124910XX relative bioavailability following ticagrelor OD tablets administered with water compared to ticagrelor IR tablets; Test type: Superiority or Other; Geometric mean ratio = 89.84, 95% CI 2-sided [82.03 to 98.39]
Statistical Analysis 5: Comparison: Treatment B vs Treatment D; Statistical assessment of metabolite AR-C124910XX relative bioavailability following ticagrelor OD tablets administered without water compared to ticagrelor IR tablets; Test type: Superiority or Other; Geometric mean ratio = 97.45, 95% CI 2-sided [90.53 to 104.90]
Statistical Analysis 6: Comparison: Treatment C vs Treatment D; Statistical assessment of metabolite AR-C124910XX relative bioavailability following ticagrelor OD tablets suspended in water and administered through NG tube compared to ticagrelor IR tablets; Test type: Superiority or Other; Geometric mean ratio = 97.07, 95% CI 2-sided [90.83 to 103.74]

2. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Time of Last Quantifiable Analyte Concentration (AUC[0-t]) of Ticagrelor and Its Active Metabolite AR-C124910XX.
Description: as for outcome 1
Time Frame: 0 hours (pre-dose) and post-dose at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36 and 48 hours in each treatment period.
Population: The PK analysis set consisted of all participants in the safety analysis set for whom at least one of the primary PK parameters, for a given analyte, can be calculated for at least two treatment periods and who had no major protocol deviations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h·ng/mL
Groups:
- Treatment C: Participants received Ticagrelor OD tablets suspended in water to be administered through a NG tube into the stomach (total of 200 mL of water).
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 30 | 31 | 33 | 33
h·ng/mL
  Ticagrelor | 3023 (28.6) | 3172 (42.6) | 3174 (40.9) | 3358 (40.0)
  AR-C124910XX | 1087 (19.7) | 1104 (20.7) | 1101 (24.4) | 1140 (23.0)
Statistical Analysis 1: Comparison: Treatment A vs Treatment D; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Geometric mean ratio = 95.04, 95% CI 2-sided [90.33 to 99.99]
Statistical Analysis 2: Comparison: Treatment B vs Treatment D; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; Geometric mean ratio = 95.41, 95% CI 2-sided [89.94 to 101.21]
Statistical Analysis 3: Comparison: Treatment C vs Treatment D; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; Geometric mean ratio = 94.66, 95% CI 2-sided [90.53 to 98.98]
Statistical Analysis 4: Comparison: Treatment A vs Treatment D; [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; Geometric mean ratio = 94.67, 95% CI 2-sided [90.94 to 98.56]
Statistical Analysis 5: Comparison: Treatment B vs Treatment D; [analysis description as in outcome 1, analysis 5]; Test type: Superiority or Other; Geometric mean ratio = 96.00, 95% CI 2-sided [91.87 to 100.33]
Statistical Analysis 6: Comparison: Treatment C vs Treatment D; [analysis description as in outcome 1, analysis 6]; Test type: Superiority or Other; Geometric mean ratio = 96.56, 95% CI 2-sided [93.08 to 100.17]

3. Primary Outcome: Area Under Plasma Concentration-time Curve From Zero to Infinity (AUC [0-∞]).
Description: as for outcome 1
Time Frame: 0 hours (pre-dose) and post-dose at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36 and 48 hours in each treatment period.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h·ng/mL
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 30 | 31 | 33 | 33
h·ng/mL
  Ticagrelor | 3068 (29.2) | 3228 (44.2) | 3226 (42.9) | 3423 (41.8)
  AR-C124910XX | 1138 (19.1) | 1155 (20.7) | 1154 (23.6) | 1197 (22.5)
Statistical Analysis 1: Comparison: Treatment A vs Treatment D; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Geometric mean ratio = 94.96, 95% CI 2-sided [90.27 to 99.89]
Statistical Analysis 2: Comparison: Treatment B vs Treatment D; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; Geometric mean ratio = 95.24, 95% CI 2-sided [89.81 to 100.99]
Statistical Analysis 3: Comparison: Treatment C vs Treatment D; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; Geometric mean ratio = 94.40, 95% CI 2-sided [90.26 to 98.73]
Statistical Analysis 4: Comparison: Treatment A vs Treatment D; [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; Geometric mean ratio = 94.82, 95% CI 2-sided [91.36 to 98.42]
Statistical Analysis 5: Comparison: Treatment B vs Treatment D; [analysis description as in outcome 1, analysis 5]; Test type: Superiority or Other; Geometric mean ratio = 95.71, 95% CI 2-sided [91.78 to 99.82]
Statistical Analysis 6: Comparison: Treatment C vs Treatment D; [analysis description as in outcome 1, analysis 6]; Test type: Superiority or Other; Geometric mean ratio = 96.50, 95% CI 2-sided [93.26 to 99.87]

4. Secondary Outcome: Time to Reach Maximum Observed Concentration (Tmax) of Ticagrelor and Its Active Metabolite AR-C124910XX.
Description: as for outcome 1
Time Frame: 0 hours (pre-dose) and post-dose at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36 and 48 hours in each treatment period.
Population: as for outcome 2
Measure: Median (Full Range); unit: h
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 30 | 31 | 33 | 33
h
  Ticagrelor | 2.02 [1.00 to 4.02] | 2.00 [1.00 to 4.00] | 2.00 [0.98 to 4.00] | 2.00 [0.98 to 4.00]
  AR-C124910XX | 3.00 [1.98 to 6.00] | 3.00 [1.98 to 4.00] | 2.00 [1.98 to 4.02] | 2.00 [1.98 to 4.00]

5. Secondary Outcome: Half-life Associated With Terminal Slope (λz) of a Semi-logarithmic Concentration-time Curve (t½λz) of Ticagrelor and Its Active Metabolite AR-C124910XX.
Description: as for outcome 1
Time Frame: 0 hours (pre-dose) and post-dose at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36 and 48 hours in each treatment period.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 30 | 31 | 33 | 33
h
  Ticagrelor | 8.02 (1.25) [1.00 to 4.02] | 8.21 (1.46) [1.00 to 4.00] | 7.99 (1.83) [0.98 to 4.00] | 8.18 (1.71) [0.98 to 4.00]
  AR-C124910XX | 9.48 (1.43) [1.98 to 6.00] | 9.35 (1.81) [1.98 to 4.00] | 9.36 (2.18) [1.98 to 4.02] | 9.47 (2.02) [1.98 to 4.00]

6. Secondary Outcome: Ratio of Metabolite Cmax to Parent Cmax, Adjusted for Differences in Molecular Weights (MRCmax) of Metabolite AR-C124910XX.
Description: Assesssment of MRCmax (ratio of metabolite Cmax to parent Cmax, adjusted for differences in molecular weights) of ticagrelor and its active metabolite AR-C124910XX following single doses of the OD tablet when administered with water, without water and suspended in water to be administered through nasogastric tubes, compared to ticagrelor IR tablets.
Time Frame: 0 hours (pre-dose) and post-dose at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36 and 48 hours in each treatment period.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 30 | 31 | 33 | 33
ratio | 0.300 (27.5) [1.98 to 6.00] | 0.277 (40.1) [1.98 to 4.00] | 0.286 (33.3) [1.98 to 4.02] | 0.271 (32.6) [1.98 to 4.00]

7. Secondary Outcome: Ratio of Metabolite AUC(0-t) to Parent AUC(0-t), Adjusted for Differences in Molecular Weights (MRAUC[0-t]) of Metabolite AR-C124910XX.
Description: Assesssment of MRAUC(0-t) (Ratio of metabolite AUC(0-t) to parent AUC(0-t), adjusted for differences in molecular weights) of ticagrelor and its active metabolite AR-C124910XX following single doses of the OD tablet when administered with water, without water and suspended in water to be administered through nasogastric tubes, compared to ticagrelor IR tablets.
Time Frame: 0 hours (pre-dose) and post-dose at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36 and 48 hours in each treatment period.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 30 | 31 | 33 | 33
ratio | 0.393 (29.8) [1.98 to 6.00] | 0.380 (42.7) [1.98 to 4.00] | 0.379 (43.2) [1.98 to 4.02] | 0.371 (43.4) [1.98 to 4.00]

8. Secondary Outcome: Ratio of Metabolite AUC [0-∞] to Parent AUC [0-∞], Adjusted for Differences in Molecular Weights (MRAUC [0-∞]) of Metabolite AR-C124910XX.
Description: Assesssment of MRAUC [0-∞] (Ratio of metabolite AUC [0-∞] to parent AUC [0-∞], adjusted for differences in molecular weights) of ticagrelor and its active metabolite AR-C124910XX following single doses of the OD tablet when administered with water, without water and suspended in water to be administered through nasogastric tubes, compared to ticagrelor IR tablets.
Time Frame: 0 hours (pre-dose) and post-dose at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36 and 48 hours in each treatment period.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 30 | 31 | 33 | 33
ratio | 0.405 (30.0) [1.98 to 6.00] | 0.391 (42.4) [1.98 to 4.00] | 0.391 (42.2) [1.98 to 4.02] | 0.382 (43.1) [1.98 to 4.00]

9. Secondary Outcome: Percentage of Participants With Adverse Events (AEs).
Description: An AE is the development of an undesirable medical condition or the deterioration of a pre-existing medical condition following or during exposure to a pharmaceutical product, whether or not considered causally related to the product. The term AE is used generally to include any AE whether serious or non-serious. A serious AE (SAE) is an AE that fulfills one or more of the following criteria: results in death, is immediately life-threatening; requires in-patient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability or incapacity or substantial disruption of the ability to conduct normal life functions; is a congenital abnormality or birth defect; is an important medical event that may jeopardize the participant or may require medical intervention to prevent one of the outcomes listed above.
Time Frame: SAEs were recorded from the signing of informed consent and AEs were recorded from randomisation until the final follow-up visit.
Population: The safety analysis set included all participants who received at least one dose of ticagrelor and for whom any safety post-dose data were available.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 31 | 32 | 34 | 33
percentage of participants
  AEs | 9.7 | 15.6 | 8.8 | 6.1
  SAEs | 0 | 0 | 0 | 0

10. Secondary Outcome: Mean Change From Baseline for Vital Signs of Supine Blood Pressure (SBP) and Diastolic BP (DBP).
Description: The following variables were collected after the participants had rested in the supine position for at least 5 minutes: SBP and DBP.
Time Frame: Day 1 (2, 4 hours post-dose) and Day 2 (24 hours post-dose).
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 31 | 32 | 34 | 33
mmHg
  SBP - Day 1, 2h Post-dose | -2 (8) | -2 (7) | -1 (8) | 3 (8)
  SBP - Day 1, 4 Post-dose | 0 (9) | 1 (8) | -1 (9) | 2 (8)
  SBP - Day 2, 24h Post-dose | -2 (6) | -1 (9) | -3 (8) | 1 (10)
  DBP - Day 1, 2h Post-dose | -1 (6) | -1 (5) | -4 (6) | 0 (5)
  DBP - Day 1, 4 Post-dose | 0 (5) | -1 (4) | -3 (5) | 0 (5)
  DBP - Day 2, 24h Post-dose | 0 (6) | -3 (5) | -3 (6) | -1 (6)

11. Secondary Outcome: Mean Change From Baseline for Vital Signs in Supine Pulse Rate.
Description: Vital signs were collected after the participant has rested in the supine position for at least 5 minutes.
Time Frame: Day 1 (2, 4 hours post-dose) and Day 2 (24 hours post-dose).
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 31 | 32 | 34 | 33
bpm
  Day 1, 2h Post-dose | 0 (5) | -1 (5) | -1 (6) | 0 (5)
  Day 1, 4 Post-dose | 1 (6) | -1 (6) | -1 (7) | 2 (5)
  Day 2, 24h Post-dose | 0 (6) | 1 (7) | 1 (7) | 1 (7)

12. Secondary Outcome: Participants With Significant Findings in 12-Lead Electrocardiography (ECG).
Description: A 12-lead ECG was obtained after the participant rested in supine position for at least 10 minutes. The study physician was to judge the overall interpretation as normal or abnormal. If abnormal, it was decided as to whether or not the abnormality was clinically significant and the reason for the abnormality was recorded.
Time Frame: At screening and at follow-up.
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 31 | 32 | 34 | 33
participants | 0 (6) | 0 (7) | 0 (7) | 0 (7)

13. Secondary Outcome: Participants With Clinically Significant Findings in Hematology, Clinical Chemistry and Urinalysis.
Description: Participants were assessed through each laboratory variables for any significant abnormalities. Hematology assessments included white blood cell count, red blood cell count, hemoglobin, hematocrit, mean corpuscular volume, mean corpuscular hemoglobin and others. Clinical chemistry assessment included testing levels of sodium, potassium, urea, creatinine, albumin, calcium, glucose (fasting) and others. Urinalysis assessment included glucose, protein, blood and microscopy (if positive for blood or protein).
Time Frame: At screening, at admission on Day -1 to each treatment period and at follow-up.
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 31 | 32 | 34 | 33
participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events were recorded from the signing of the informed consent and adverse events were recorded from randomization until the final follow-up visit.
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/32 | 0/34 | 0/33
Other Adverse Events (participants affected / at risk) | 3/31 | 5/32 | 3/34 | 2/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A (N=31) | Treatment B (N=32) | Treatment C (N=34) | Treatment D (N=33)
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Thrombophlebitis (Vascular disorders) | 0 | 2 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a publication (e.g., in a scientific journal) based on the results of this study is envisaged, approval from AstraZeneca will be obtained and a draft manuscript will be submitted to AstraZeneca for scrutiny and comment. The choice of conduit will be mutually agreed on by the Principal Investigator and AstraZeneca.